CLINICAL TRIAL: NCT05023967
Title: Time Restricted Eating And Metformin (TEAM) in Invasive Breast Cancer (IBC) or Ductal Carcinoma in Situ (DCIS). A Randomized, Phase IIb, Window of Opportunity Presurgical Trial.
Brief Title: Metformin and Nightly Fasting in Women With Early Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021-0901; NCI-2021-08921 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); B115UCS2019; 2021-000134-34; 2021-09-01; Pending3 (Other: M D Anderson Cancer Center); MDA20-02-01 (Other: DCP); UG1CA242609 (NIH)
Record Dates: First submitted 2021-08-26; First posted 2021-08-27 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-11

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Breast Ductal Carcinoma In Situ; Invasive Breast Carcinoma
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating | interventions — Specimen Handling; Metformin; Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (fasting, glucose monitoring, counseling, metformin) (Experimental): Patients fast for >= 16 hours every night and use the continuous glucose monitoring system for 4-6 weeks. Patients also receive nutritional counseling sessions on days 0 and 10. Beginning week 2, patients also receive metformin hydrochloride extended release PO QD until the day of surgery. Treatment continues for 4-6 weeks (until surgery) in the absence of disease progression or unacceptable toxicity. Patients undergo the collection of blood samples at baseline and at the final study visit (days 28-43), and the collection of tissue at the time of surgery (days 28-43).
  Interventions: Procedure: Biospecimen Collection; Drug: Extended Release Metformin Hydrochloride; Other: Monitoring; Other: Nutritional Assessment; Other: Short-Term Fasting
- Arm II (glucose monitoring) (Active Comparator): Patients continue their usual dietary pattern and use the continuous glucose monitoring system for 4-6 weeks (until surgery). Patients undergo the collection of blood samples at baseline and at the final study visit (days 28-43), and the collection of tissue at the time of surgery (days 28-43).
  Interventions: Procedure: Biospecimen Collection; Other: Monitoring

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood and tissue samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Extended Release Metformin Hydrochloride — Given PO
  Other Names: ER Metformin Hydrochloride; Extended-release Metformin Hydrochloride; Glucophage XR; Glumetza; Metformin Hydrochloride Extended Release
  Arms: Arm I (fasting, glucose monitoring, counseling, metformin)
Other: Monitoring — Use continuous glucose monitoring system
  Other Names: monitor
Other: Nutritional Assessment — Receive nutritional counseling
  Other Names: Dietary Assessment; dietary counseling; nutritional counseling
  Arms: Arm I (fasting, glucose monitoring, counseling, metformin)
Other: Short-Term Fasting — Perform intermittent fasting
  Other Names: Intermittent Fasting; Short-term Intermittent Fasting
  Arms: Arm I (fasting, glucose monitoring, counseling, metformin)

SUMMARY:
This phase IIb trial studies the combined effect of prolonged nightly fasting and metformin hydrochloride extended release in decreasing breast tumor cell proliferation and other biomarkers of breast cancer. Preventing invasive breast cancer or DCIS. Metformin is widely used to treat type II diabetes and is associated with a decreased risk of cancer and death in diabetic individuals. Intermittent fasting may protect cancer patients from the toxic effects of chemotherapy agents without causing chronic weight loss. The combination of intermittent fasting and metformin may reduce breast cancer growth and may be used in women at risk for breast cancer or other cancers associated with being overweight.

DETAILED DESCRIPTION:
- Primary Interim Objective

The primary interim objective will be to assess the safety of the experimental intervention based on the frequency of occurrence of a Dose Limiting Toxicity (DLT) in the first 14 participants assigned to the experimental treatment arm. A DLT is defined as a hypoglycemic event requiring permanent discontinuation of study treatment or any grade 3 or greater adverse event (AE) possibly, probably, or definitely related to the study drug.

Hypoglycemia AEs that require permanent discontinuation of study treatment are:

* ≥ 1 grade 2 or higher neuroglycopenic symptoms and grade 2 hypoglycemia;
* occurrence ≥ 3 times of grade 2 symptoms (≥ 2 autonomic or ≥ 1 neuroglycopenic symptoms) and grade 1 or higher hypoglycemia;
* symptomatic or asymptomatic grade 3 hypoglycemia.

In the first 14 participants enrolled in the experimental arm (combination of prolonged nightly fasting and Metformin Hydrochloride Extended-Release) we can accept at most 3 participants with a DLT. If 4 or more of the first 14 participants assigned to the treatment arm experience the above-mentioned DLTs, the trial will be definitively stopped.

In order to early identify any DLT, participants will be instructed to contact study staff in case of occurrence of any symptoms regardless of their grade and a review of the occurrence of any AE will be performed every 10 days. The early detection of symptoms related to the study treatment will help us to avoid worsening of symptoms to grade 3 and thus prevent any DLT. Moreover, the glucose trends of the first 14 participants enrolled in the experimental arm will be downloaded and immediately evaluated to identify any asymptomatic hypoglycemia.

Hypoglycemia will be assessed through the evaluation of glucose reports and fingersticks results in case of symptoms.

- Primary and Co-primary Objective

We have recently shown that the combination of hypoglycemia and Metformin reduces tumor growth in animal models (1). Moreover, Metformin alone was able to reduce breast cancer cell proliferation in women with insulin resistance in a randomized presurgical trial (2,3).

Breast carcinogenesis may be present in three components in surgical specimens and more rarely in biopsy specimens: invasive breast cancer (IBC), ductal carcinoma in situ (DCIS) and intraepithelial neoplasia (IEN), defined as atypical ductal hyperplasia (ADH) or atypical lobular hyperplasia (ALH) or lobular carcinoma in situ (LCIS). We propose to assess the effect of the combination of prolonged nightly fasting (≥16 hours) and Metformin Hydrochloride Extended-Release on the change of Ki67 labeling index (LI) in cancer tissue (IBC or DCIS, if IBC is absent) between pre-treatment biopsy and post treatment surgical specimen. As co-primary objective, we will also evaluate the difference in post-treatment Ki67 LI in cancer adjacent DCIS (in the presence of IBC), if present, or IEN (defined as ADH or ALH or LCIS) between the active treatment and the control group. IBC and DCIS strata will be based on the post-treatment pathology. If DCIS is the primary lesion because of the absence of invasive disease, adjacent IEN will be counted only if ADH/ALH/LCIS is present.

The change (pre/post treatment) of Ki67 LI in IEN will be evaluated only if present in the pretreatment biopsy specimen.

Secondary Objectives

* to explore the effect of intervention on the change of expression of PP2A-GSK3ß-MCL-1 axis in pre-post treatment cancer tissue levels;
* to measure the change in circulating biomarkers: HOMA index, Hb1Ac;
* to measure the difference of cell death by IHC for M30 in post- treatment cancer samples between arms;
* to measure the difference of pS6 by IHC in post- treatment cancer samples between arms;
* to compare the area under the curve (AUC) of glucose levels between arms according to insulin resistance biomarker levels and WCRF score;
* to assess safety and toxicities according to NCI-CTC AE v. 5.0.
* Exploratory Objectives
* to correlate a customized NGS mutational profile panel focused on ER+ve with the response of Ki67;
* to measure the change in circulating biomarkers: highly sensitive CRP (hsCRP), C-peptide, IGF-I, IGFBP-1, IGFBP-3, free IGF-I, lipid profile, adipokines (leptin and adiponectin);
* to correlate psychological distress, eating habits, tobacco and alcohol consumption with the response of Ki67 and insulin resistance biomarkers between arms;
* to compare the slow ramp up schedule of metformin to the quick ramp up schedule to metformin in the treatment group on the area under the curve (AUC) of glucose levels

ELIGIBILITY:
Inclusion Criteria:

* Women with histologically confirmed luminal (ER+ve and/or progesterone [PgR]+ve >= 1%) operable IBC (cT1-2, cN0-1, Mx) candidate to elective surgery and not to neo-adjuvant treatment. Women with larger tumors who refuse neo-adjuvant chemotherapy before surgery can also be eligible. Luminal HER2+ve (cT1, cN0) IBC and DCIS are also eligible
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Leukocytes >= 3,000/microliter
* Absolute neutrophil count >= 1,500/microliter
* Platelets >= 100,000/microliter
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 1.5 x institutional upper limit of normal
* Creatinine within normal institutional limits
* Creatinine clearance estimated with Cockcroft-Gault formula > 45 mL/min
* Female participants of child-bearing potential must agree to use contraception such as barrier method of birth control or abstinence, prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she has to inform her study physician immediately. The effects of metformin hydrochloride extended release on the developing human fetus at the recommended therapeutic dose are unknown
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Body mass index (BMI) < 18.5 Kg/m^2
* Previous treatment for breast cancer including chemotherapy and endocrine therapy within the last 12 months
* Women who are planned to receive neoadjuvant therapy
* Triple negative breast cancer (BC)
* Patients with a history of cancer within the last year. NOTE: Non melanoma skin cancer is allowed.
* Documented history of symptomatic hypoglycemia
* Diabetic patients or participants with fasting glucose level >= 126 mg/dL
* Known hypersensitivity or intolerance to metformin hydrochloride extended release
* Participants should not be receiving any other investigational agents
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* History of lactic acidosis
* Liver dysfunction including chronic active hepatitis and cirrhosis not compensated
* History of vitamin B12 deficiency or megaloblastic anemia
* Chronic use of large doses of diuretics (e.g., > 80 mg furosemide)
* Current use of oral hormonal contraceptives or female hormones in the last four weeks or 5 half-lives, excluding vaginal creams and intrauterine devices (IUDs)
* Concomitant use of topiramate or other carbonic anhydrase inhibitors (e.g., zonisamide, acetazolamide or dichlorphenamide)
* Pregnant or lactating women. Pregnant women are excluded from this study because even though published data from post-marketing studies have not reported a clear association between metformin hydrochloride extended release and major birth defects, miscarriage, or adverse maternal or fetal outcomes when metformin hydrochloride extended release was used during pregnancy, these studies cannot definitely establish the absence of any metformin hydrochloride extended release associated risk because of methodological limitations, including small sample size and inconsistent comparator groups. Because there is an unknown but potential risk for adverse events (AEs) in nursing infants secondary to treatment of the mother with metformin hydrochloride extended release, breastfeeding should be discontinued if the mother is treated with metformin hydrochloride extended release. Moreover, prolonged fasting is not recommended in pregnant woman
* Women who practice any type of intermittent fasting program
* Women who will not have anyone available to assist them in case of need

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2025-12-09 (Actual); Study Completion 2026-12-16 (Estimated)

PRIMARY OUTCOMES:
Frequency of occurrence of dose limiting toxicity | Up to 4-6 weeks
  Defined as a hypoglycemic event requiring permanent discontinuation of study treatment or any grade 3 or greater adverse event possibly, probably, or definitely related to the study drug.
Change in pre-post treatment Ki67 labeling index in invasive breast cancer (IBC) or ductal carcinoma in situ (DCIS) (in the absence of IBC) | Baseline up to 4-6 weeks
  Generalized linear models will be used to assess differences between treatment arms for Ki67. Log transformation will be considered to obtain normal distribution of residuals. Will also evaluate the need to adjust for baseline characteristics and significant confounders (such as body mass index [BMI] and HER2 status).
Difference in post-treatment adjacent DCIS (in the presence of IBC), if present, or intraepithelial neoplasia Ki67 between arms | Post-treatment (4-6 weeks)
  Generalized linear models will be used to assess differences between treatment arms for Ki67. Log transformation will be considered to obtain normal distribution of residuals. Will also evaluate the need to adjust for baseline characteristics and significant confounders (such as BMI and HER2 status).

SECONDARY OUTCOMES:
Change in circulating biomarkers | Baseline up to 4-6 weeks
  Will include Homeostatic model assessment index, highly sensitive C-reactive protein, C-peptide, IGF-I, IGFBP-1, IGFBP-3, free IGF-I, Hb1Ac, lipid profile, leptin and adiponectin. Will present full distributions and median values of circulating biomarkers, Ki67, at baseline, after treatment, and of changes and percentage changes (with interquartile ranges) of all continuous variables, by arms. Analysis of covariance (ANCOVA) models will evaluate the associations of post values (after treatment) and changes from baseline by study arms adjusting for baseline values, explanatory variables and possible confounders (such as age and BMI). Normal distribution of residuals from full models will be checked and, if needed, a transformation will be considered.
Change of CIP2A-PP2A-GSK3beta-MCL-1 axis in cancer tissue | Baseline up to 4-6 weeks
  Will present full distributions and median values of circulating biomarkers, Ki67, at baseline, after treatment, and of changes and percentage changes (with interquartile ranges) of all continuous variables, by arms. ANCOVA models will evaluate the associations of post values (after treatment) and changes from baseline by study arms adjusting for baseline values, explanatory variables and possible confounders (such as age and BMI). Normal distribution of residuals from full models will be checked and, if needed, a transformation will be considered.
Change of Ki67 in cancer tissue | Baseline up to 4-6 weeks
  Will depend upon next generation sequencing mutational profile obtained in post-treatment surgical specimens. Will present full distributions and median values of circulating biomarkers, Ki67, at baseline, after treatment, and of changes and percentage changes (with interquartile ranges) of all continuous variables, by arms. ANCOVA models will evaluate the associations of post values (after treatment) and changes from baseline by study arms adjusting for baseline values, explanatory variables and possible confounders (such as age and BMI). Normal distribution of residuals from full models will be checked and, if needed, a transformation will be considered.
Difference of M30 | Post-treatment
  Will be assessed between arms. Will be assessed using IHC.
Difference of phosphorylated S6 | Post-treatment
  Will be assessed between arms. Will be assessed using IHC.
Physiological distress | Up to 4-6 weeks
  Will be correlated with response biomarkers.
Eating habits | Up to 4-6 weeks
  Will be correlated with response biomarkers.
Tobacco | Up to 4-6 weeks
  Will be correlated with response biomarkers.
Alcohol consumption | Up to 4-6 weeks
  Will be correlated with response biomarkers.
Incidence of adverse events | Up to 4-6 weeks
  Evaluated according to the Common Terminology Criteria for Adverse Events version 5.0.
Difference of the area under the curve of glucose levels | Up to 4-6 weeks
  Will be assessed between arms.

CONTACTS AND LOCATIONS:
Overall Officials: Parijatham Thomas, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- M D Anderson Cancer Center, Houston, Texas, United States
- Italy (2):
  - Galliera Hospital, Genoa
  - European Institute of Oncology, Milan

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm